CLINICAL TRIAL: NCT04297800
Title: Gait Characteristics and Cognitive Evolution in Parkinson Disease (GECO-PARKINSON STUDY)
Brief Title: Gait Characteristics and Cognitive Evolution in Parkinson Disease
Acronym: GECO-PD
Status: Completed | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: GECO-PARKINSON STUDY
Record Dates: First submitted 2020-01-20; First posted 2020-03-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease
Keywords: gait; attention/executive function domain; device; walk parameters; wireless inertial sensor
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Parkinson's disease (PD) is a chronic progressive nervous system disease with gradual motor impairment. Cognitive dysfunction is common in PD, even in the early stages, and it is characterized by impairments in executive, attention, memory, language and visuospatial function. Motor symptoms, in particular, alterations in gait, have been studied in clinical practice to assess disease progression, and its response to treatments, both farmacological and physiotherapeutic.

Recent research on wearable technology in PD has shown that motor tests can be automated using wearable technology to eliminate human supervision and patient-reported data. Particularly, the quantitative gait analysis by using inertial devices has been proposed as a sensitive tool to longitudinally monitor gait worsening, response to dopaminergic treatment over time and cognitive dysfunction in PD patients.

The aim of this prospective multicente observational study is to investigate whether the dysfunction of specific gait parameters may be correlated to cognitive impairment (Attention/Executive Function Domain) in a cohort of ambulatory PD patients followed for 3 years.

DETAILED DESCRIPTION:
This is a prospective multicenter observational study with annual follow-up assessments over 3 years.

Gait is assessed by an inertial device (BTS G-WALK). G- WALK is an easy-to-use solution to obtain accurate, objective and quantitative spatial-temporal gait data. The device is a wireless system consisting of an inertial sensor composed by a triaxial accelerometer, a magnetic sensor, and a triaxial gyroscope that positioned on lumbar/ or sacral segments allows a functional gait analysis.

Cognitive performance is evaluated with a neuropsychological battery designed to assess memory, executive /attention, and visuospatial domains.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Aged between 55-74 years
* Diagnosis of idiopathic PD based on MDS clinical diagnostic criteria
* Hoehn & Yahr (H&Y) stages 2 to 3 at enrollment, independently by PD duration
* Clinical-pharmacological stabilization until 3 months before the enrollment
* DBS treatment (stable stimulation parameters until 6 months before the enrollment)

Exclusion Criteria:

* Evidence of neurodegenerative and secondary parkinsonism
* Dementia ( (score <25 on the Mini Mental State Examination - MMSE)
* Psychiatric disorder (Beck Depression Inventory-II - BDI-II Score >19)
* Presence of organ failure (Modified Cumulative Illness Rating Scale - CIRS > 2)
* Orthopedic disorder or co-morbidities that may affect gait
* Drug and alcohol use

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-11-09 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Gait assessed by 6-Minute Walk Test (6MWT) | Every year for 3 years
  Gait assessment
Changes in Gait assessed by Extended-Time Up and Go (eTUG) | Every year for 3 years
  Gait assessment
Changes in cognitive function assessed by Mini-Mental State Examination (MMSE) | Every year for 3 years
  Cognitive Assessment. The MMSE score ranges from 0 to 30 points, in which a lower score indicates a higher degree of cognitive impairment.
Changes in cognitive function assessed by the Montreal Cognitive Assessment (MoCA) | Every year for 3 years
  Cognitive Assessment. The total score of the MoCA is 30 points, with a score less than 24 is considered cognitive impairment.
Changes in cognitive function assessed by Frontal Assessment Battery (FAB) | Every year for 3 years
  Cognitive Assessment

SECONDARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale, part III | Every year for 3 years
  The MDS-UPDRS III is the sum of 33 scores that evaluate Parkinson's disease motor symptoms on a scale from 0 to 4 points. The total scale range is 0-132, where higher scores indicate more severe symptoms.
"Rapid eye movement Sleep" Behavior Disorder Screening Questionnaire | Every year for 3 years
  The RBDSQ ranges from 0 to 13, where higher scores represent a worse outcome.
Hyposmia Rating Scale | Every year for 3 years
  The scale ranges from 6 to 24, where higer scores indicate more worse sense of olfaction.
short Falls Efficacy Scale | Every year for 3 years
  s-FES ranges from 7 to 28, where higher scores indicate high level of concern about falling during social and physical activities inside and outside the home.
Berg Balance Scale | Every year for 3 years
  The BBC includes 14 functional balance. The scale ranges from 0 to 56, where higer scores indicate that the participant can complete the tasks.
Tinetti test | Every year for 3 years
  The test grants a maximum of 16 points for static part (sitting) and 12 point for dynamic (walking) part. Higher is the score, better is the performance
Parkinson's Disease Questionnaire | Every year for 3 years
  PDQ-8 ranges from 0 to 32, where higher scores reflect a lower health-related quality of life.
Beck Anxiety Index | Every year for 3 years
  The BAI range is 0- 63, where higer scores indicate more severe symptoms.
Beck Depression Inventory II | Every year for 3 years
  The BDI-II ranges from 0 to 63, where higer scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dario Alimonti, MD, PhD, Principal Investigator — ASST- Papa Giovanni XXIII; Francesco Biroli, MD, Study Chair — Fondazione per la Ricerca Ospedale di Bergamo (FROM)
Locations (3):
- Italy (3):
  - ASST- Papa Giovanni XXIII, Bergamo
  - Spedali Civili di Brescia, Brescia
  - Ospedale San Gerardo di Monza, Monza